CLINICAL TRIAL: NCT05922254
Title: Combined Effects of Active Cycle of Breathing Technique and Autogenic Drainage in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Combined Effects of ACBT and AUTOGENIC DRAINAGE in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0318
Record Dates: First submitted 2023-06-06; First posted 2023-06-28 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive; Drainage; Postural; Pulmonary Disease; Respiratory Therapy.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active cycle of breathing technique (Active Comparator): Group A is a control group. First, the patients will receive baseline treatment (pursed lip breathing). Additionally, patients will be administered the Active Cycle of Breathing Technique after receiving the Baseline Treatment
  Interventions: Other: Active cycle of breathing technique
- Autogenic drainage (Experimental): Both the physiotherapist's hand and the subject's hands were put on the subject's abdomen to feel the activity of the abdominal muscles. The patient inhaled slowly through the nose while using their diaphragm and holding their breath for two to three seconds to allow collateral ventilation to bring air behind their secretions. Exhalation was done through the mouth. The palm of the therapist placed on the upper chest felt the vibration of the mucous. Their positions were disclosed by the vibrations' frequency. Secretions in tiny airways can be seen using high frequencies. The method has phases for unsticking, collecting and evacuation. The mucus was expelled by a stronger expiration or a high lung volume huff at the conclusion of the session.
  Interventions: Other: Active cycle of breathing technique; Other: Autogenic drainage

INTERVENTIONS:
Other: Active cycle of breathing technique — The ACBT technique consists of three different breathing techniques: breathing control, thoracic expansion exercises and forced expiration technique. 1. Breathing Control 2. Thoracic Expansion Exercises: 3. Forced Expiration Technique:
Other: Autogenic drainage — Huffing or blowing the nose helped to get rid of any secretions in the upper airways. The therapist was placed close enough to hear the subject's breathing while sitting to the side and slightly behind the patient. Both the physiotherapist's hand and the subject's hands were put on the subject's abdomen to feel the activity of the abdominal muscles. The patient inhaled slowly through the nose while using their diaphragm and holding their breath for two to three seconds to allow collateral ventilation to bring air behind their secretions. Exhalation was done through the mouth. The palm of the therapist placed on the upper chest felt the vibration of the mucous. Their positions were disclosed by the vibrations' frequency.
  Arms: Autogenic drainage

SUMMARY:
A randomised controlled trial will be conducted with COPD patients as its target population. There will be 40 individuals for both the control group and the intervention group. Group A is a control group while Group B is an experimental group (20 participants on Group A and 20 on group B). The baseline treatment for both groups were pursed lip breathing and ACBT. On the other hand, group B experimental group will also undergo (pursued lip breathing and ACBT) with autogenic drainage. Group A session lasts for 30 minutes and Group B session lasts for 45 minutes. There is only one session per day. There is a three session in a week for 4 weeks. Measurements are made of dyspnea, oxygen saturation, peak expiratory flow rate, pulse rate and fatigue both before and after the treatment, data were recorded. Participants in the trial must have mild to moderate COPD (GOLD Criteria) and be between the ages of 40 to 60 years. Data from Sheikh Zayed Hospital, Rahim Yar Khan will be collected. Follow-up for both completed tasks and changes in pulmonary status will be evaluated after 4 weeks. Modified Borg Dyspnea (RPE) Scale, Breathlessness, Cough and Sputum Scale (BCSS), Fatigue Severity Scale or Visual Analogue Scale, Peak flow meter, Oximeter will be used to measure the outcomes. Data will be analysed using the SPSS 21.0 Statistical Software

DETAILED DESCRIPTION:
The term "COPD" refers to a range of illnesses that impair breathing and obstruct airflow.

Smoking or having smoked in the past increases the risk of developing COPD because tobacco smoke is the primary cause of the disease. The risk is further increased by family history, occupational or home, air pollution exposure and respiratory illnesses including pneumonia. The signs and symptoms include wheezing, coughing up mucus (sputum) and difficulty in breathing. It is frequently brought on by prolonged exposure to irritant gases or particulates most frequently from cigarette smoke. Heart disease, lung cancer and a number of other diseases are more likely to occur in people with COPD.

A randomised controlled trial will be conducted with COPD patients as its target population. There will be 40 individuals for both the control group and the intervention group. Group A is a control group while Group B is an experimental group (20 participants on Group A and 20 on group B). The baseline treatment for both groups were pursed lip breathing and ACBT. On the other hand, group B experimental group will also undergo (pursued lip breathing and ACBT) with autogenic drainage. Group A session lasts for 30 minutes and Group B session lasts for 45 minutes. There is only one session per day. There is a three session in a week for 4 weeks. Measurements are made of dyspnea, oxygen saturation, peak expiratory flow rate, pulse rate and fatigue both before and after the treatment, data were recorded. Participants in the trial must have mild to moderate COPD (GOLD Criteria) and be between the ages of 40 to 60 years. Data from Sheikh Zayed Hospital, Rahim Yar Khan will be collected. Follow-up for both completed tasks and changes in pulmonary status will be evaluated after 4 weeks. Modified Borg Dyspnea (RPE) Scale, Breathlessness, Cough and Sputum Scale (BCSS), Fatigue Severity Scale or Visual Analogue Scale, Peak flow meter, Oximeter will be used to measure the outcomes. Data will be analysed using the SPSS 21.0 Statistical Software.

ELIGIBILITY:
Inclusion Criteria:

* Both genders (Male and Female)
* Age 40 to 60 years
* Mild to moderate COPD (According to GOLD Criteria)
* Patient is bilingual.

Exclusion Criteria:

* Patients having progressive respiratory muscle weakness (Mysthenia Gravis)
* Cardiovascular impairment
* Any recent surgery
* Systemic illness
* Angina
* Uncontrolled diabetes and hypertension
* TB
* Non-cooperative Patients

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Modified Borg Dyspnea (RPE) scale | fourth week
  The most popular tool for evaluating symptoms of breathlessness is the Modified Borg Dyspnoea Scale. RPE scales, despite being a subjective gauge of exercise intensity, are useful when utilised properly. The RPE scale has a 0 to10 scale with 0 being no exertion and 10 being maximum effort
Dyspnea Index Questionnaire | fourth week
  The Dyspnoea Index questionnaire is a useful tool for quantifying upper airway dyspnea symptoms in patients. It includes 10-item surveys
Breathlessness, Cough and Sputum Scale (BCSS) | fourth week
  The breathlessness, cough and sputum scale (BCSS) are a three-item scale that rates symptoms of dyspnea, cough and sputum on a Likert scale from 0 (no symptoms) to 4 (severe symptoms). The Breathlessness, Cough and Sputum Scale (BCSS), which assesses common symptoms found in the COPD population, is used to predict patient exacerbations
Fatigue Severity Scale | fourth week
  You can assess the impact of fatigue on you using the Fatigue Severity Scale (FSS). The FSS is a brief questionnaire that asks you to rate how tired you are. Nine statements in the FSS questionnaire allow you to express how severe your tiredness symptoms are
Peak Flow meter | baseline and fourth week
  A peak flow meter must be used by blowing forcefully into it. In liters per minute, the meter measures the forced air flow. When you exhale, the indicator on the device moves and gives you a reading on a scale of 1 to 10. When a person's airway function changes, it may be a sign that their asthma or COPD symptoms are getting worse. This is where a peak flow meter is useful
Oximeter | fourth week
  The oxygen saturation level of your blood can be measured with a non-invasive procedure called pulse oximetry. It can quickly identify even minute variations in oxygen levels. These levels demonstrate how well blood transports oxygen to your arms and legs, which are the extremities that are farthest from your heart. It looks like a little clip and is called a pulse oximeter. It attaches to a body component, usually a finger

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Sheikh Zayed Hospital,, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yadav UN, Lloyd J, Hosseinzadeh H, Baral KP, Harris MF. Do Chronic Obstructive Pulmonary Diseases (COPD) Self-Management Interventions Consider Health Literacy and Patient Activation? A Systematic Review. J Clin Med. 2020 Feb 28;9(3):646. doi: 10.3390/jcm9030646. PMID 32121180
- [Background] Garcia-Aymerich J, Lange P, Benet M, Schnohr P, Anto JM. Regular physical activity reduces hospital admission and mortality in chronic obstructive pulmonary disease: a population based cohort study. Thorax. 2006 Sep;61(9):772-8. doi: 10.1136/thx.2006.060145. Epub 2006 May 31. PMID 16738033
- [Background] Mendes LP, Moraes KS, Hoffman M, Vieira DS, Ribeiro-Samora GA, Lage SM, Britto RR, Parreira VF. Effects of Diaphragmatic Breathing With and Without Pursed-Lips Breathing in Subjects With COPD. Respir Care. 2019 Feb;64(2):136-144. doi: 10.4187/respcare.06319. Epub 2018 Aug 28. PMID 30154127